CLINICAL TRIAL: NCT02128399
Title: Antimicrobial Stewardship Reduces MDRO Isolates in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Jianfeng Xie (Other)
Responsible Party: Sponsor-Investigator, Jianfeng Xie, doctor of department of critical care medicine, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: MDRO
Record Dates: First submitted 2014-04-22; First posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2012-07

CONDITIONS: Sepsis
Keywords: antimicrobial stewardship
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- patients before and after intervetion

SUMMARY:
Antimicrobial exposure is known to reduce the selection for various drug-resistant organisms. Numerous studies have demonstrated the association between antimicrobial use and MDR bacteria detection. However, to the investigators knowledge, there is few data to support the concept that reducing antibiotic use actually leads to improvements in antibiotic susceptibilities. Moreover, antimicrobial stewardship was demonstrated to reduce MDRO and was strongly recommended in clinics. As the investigators know, antimicrobial overuse, which occurs commonly in China, induces a severe antibacterial resistance. China's Ministry of Health (MOH) has established a policy about the antimicrobial stewardship. To date, the investigators do not have published documentation the effects of this policy on multidrug-resistant organism (MDRO) in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the ICU

Exclusion Criteria:

* Patients who were readmitted to the ICU during a single hospital stay

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients who admitted into intensive care unit
Sampling Method: Probability Sample
Enrollment: 978 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The number of participates infection or colonization with MDRO in critically ill patients at ICU admission and discharge as a measure of effect of antimicrobial stewardship | up to 90 days
  MDRO isolation from inclusion to the date of discharge of hospital, access up to 90 days

REFERENCES:
- [Derived] Ma X, Xie J, Yang Y, Guo F, Gao Z, Shao H, Huang Y, Yang C, Qiu H. Antimicrobial stewardship of Chinese ministry of health reduces multidrug-resistant organism isolates in critically ill patients: a pre-post study from a single center. BMC Infect Dis. 2016 Nov 25;16(1):704. doi: 10.1186/s12879-016-2051-8. PMID 27887595